CLINICAL TRIAL: NCT00740792
Title: Randomized, Double-Blind Trial of MP29-02 Nasal Spray Compared to Placebo, Azelastine Hydrochloride Nasal Spray, and Fluticasone Propionate Nasal Spray in the Treatment of Patients With Seasonal Allergic Rhinitis.
Brief Title: A Study Evaluating the Safety and Effectiveness of a Nasal Spray to Treat Seasonal Allergies
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Meda Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MP4004
Record Dates: First submitted 2008-08-22; First posted 2008-08-25 (Estimated); Results first posted 2012-09-07 (Estimated); Last update posted 2012-09-07 (Estimated); Status verified 2012-08

CONDITIONS: Seasonal Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal | interventions — MP29-02; azelastine; Fluticasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- azelastine HCl/fluticasone propionate (Experimental): nasal spray
  Interventions: Drug: azelastine HCl/fluticasone propionate
- azelastine HCL (Active Comparator): nasal spray
  Interventions: Drug: azelastine Hcl
- fluticasone propionate (Active Comparator): nasal spray
  Interventions: Drug: fluticasone propionate
- placebo (Placebo Comparator): nasal spray
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: azelastine HCl/fluticasone propionate — azelastine HCl 548 mcg/ fluticasone propionate 200 mcg one spray per nostril BID
  Other Names: MP29-02
  Arms: azelastine HCl/fluticasone propionate
Drug: azelastine Hcl — azelastine Hcl 548 mcg one spray per nostril BID
  Other Names: azelastine hydrochloride
  Arms: azelastine HCL
Drug: fluticasone propionate — fluticasone propionate 200 mcg one spray per nostril BID
  Arms: fluticasone propionate
Drug: placebo — placebo one spray per nostril BID
  Arms: placebo

SUMMARY:
The purpose of this study is to determine if two allergy medications (formulated azelastine and fluticasone product) are more effective than placebo or either medication alone (azelastine or fluticasone)

DETAILED DESCRIPTION:
This will be a Phase III, randomized, double-blind, placebo-controlled, parallel-group study in subjects with moderate-to-severe seasonal allergic rhinitis (SAR). The study will begin with a 7-day, single-blind, placebo lead-in period (Day -7 to Day 1). Subjects will be instructed to take placebo lead-in medication twice daily (1 spray per nostril), approximately every 12 hours. On Day 1, subjects who satisfy the symptom severity requirements and continue to meet all of the study inclusion/exclusion criteria will be randomized in a 1:1:1:1 ratio to receive 1 spray per nostril twice daily of MP29-02, azelastine hydrochloride, fluticasone propionate, or placebo nasal spray.

Efficacy will be assessed by the change from baseline in the subject-reported 12-hour reflective Total Nasal Symptom Score (TNSS). On Days 1 through 14, subjects will rate the instantaneous and reflective TNSS symptoms of sneezing, nasal congestion, runny nose, and nasal itching; the instantaneous and reflective total ocular symptom score (TOSS) symptoms of itchy eyes, watery eyes and eye redness; the symptom of postnasal drip will be rated, reflectively, twice daily (AM and PM) in a diary prior to the dose of study medication. Symptoms will be scored on a 0 to 3 scale (0 = no symptoms, 1 = mild symptoms, 2 = moderate symptoms, 3 = severe symptoms), such that the maximum daily symptom severity score will be 24 for the TNSS and 18 for the TOSS. Additional secondary efficacy variables will include reflective individual nasal and ocular symptom scores, as well as change from Baseline to Day 14 in the Rhinoconjunctivitis Quality of Life Questionnaire (RQLQ).

Subjects ≥ 18 years of age will complete the RQLQ on Day 1 (prior to dosing) and Day 14. Subjects will return to the clinic on Day 7 for an interim evaluation. After completing the 2-week double-blind treatment period, subjects will return to the clinic on Day 14 (or at time of early termination) for an end-of-study evaluation. Safety and tolerability assessments will be made on Days 7 and 14. Tolerability will be evaluated by subject-reported adverse events (AEs), nasal examinations, and vital signs assessments.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects 12 years of age and older
* Provide written informed consent/pediatric assent. If the subject is a minor, parent or legal guardian must give written informed consent
* Subjects must have moderate-to-severe rhinitis, defined as having one or more of the following:

  1. Sleep disturbance
  2. Impairment of daily activities, leisure and/or sport
  3. Impairment of school or work
  4. Troublesome symptoms
* Screening Visit: Have a 12-hour reflective TNSS of at least 8 of 12 and a congestion score of 2 or 3 on Visit 1
* Randomization Visit: Have a 12-hour reflective TNSS (AM or PM) of at least 8 on 3 separate symptom assessments (one of which was within 2 days of Day 1, and can include the morning of Day 1) during the Lead-in Period.
* Randomization Visit: Have an AM or PM 12-hour reflective nasal congestion score of 2 or 3 must have been recorded on 3 separate symptom assessments (one of which was within 2 days of Day 1, and can include the morning of Day 1) Randomization Visit: Have an instantaneous TNSS score of 8 or more at time point zero, just prior to beginning the onset of action assessment
* Have taken at least 10 doses of the lead-in medication
* Willing and able to comply with the study requirementsAt least a 2-year history of SAR during Fall allergy season
* The presence of IgE-mediated hypersensitivity to a local Fall pollen, confirmed by a positive response to skin prick within the last year. A positive response is defined as a wheal diameter of at least 3 mm larger than the negative control.
* General good health and free of disease or concomitant treatment that could interfere with the interpretation of the study results
* Subjects receiving immunotherapy injections (antigen desensitization) must be on a stable maintenance regimen for at least 30 days before the first study visit
* Subjects currently receiving sublingual immunotherapy are excluded. A 6-month washout period is required following the last dose of sublingual immunotherapy.

Exclusion Criteria:

* On Focused Nasal Examination, the presence of any superficial and moderate nasal mucosal erosion, nasal mucosal ulceration, or nasal septum perforation at either the screening visit or randomization visit
* Other nasal disease(s) likely to affect deposition of intranasal medication
* Nasal surgery or sinus surgery within the previous year.
* Chronic sinusitis - more than 3 episodes per year
* Planned travel outside of the pollen area during the study period
* The use of any investigational drug within 30 days prior to Day -7.
* Presence of any hypersensitivity to drugs similar to azelastine hydrochloride or fluticasone propionate
* Women who are pregnant or nursing
* Women of childbearing potential who are not abstinent or not practicing a medically acceptable method of contraception*
* Respiratory Tract Infections within 14 days prior to Day -7
* Respiratory Tract Infections requiring antibiotic treatment 14 days prior to Day -7
* Asthma (with the exception of intermittent asthma).
* Significant pulmonary disease including COPD
* Clinically significant arrhythmia or symptomatic cardiac conditions
* A known history of alcohol or drug abuse within the last 2 years
* Existence of any surgical or medical condition or physical or laboratory findings that could interfere with study result interpretation.
* Patients with a history of Glaucoma
* Clinically relevant abnormal physical findings within 1 week of randomization that may preclude compliance with the study procedures
* Employees of the research center or private practice and their family members are excluded
* Subjects who participated in protocol MP4001 or MP4002

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 776 (Actual)
Dates: Start 2008-08; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lewis M Fredane, MD, Study Director — Meda Pharmaceuticals
Locations (39):
- United States (39):
  - Allergy, Asthma and Immunology Associates, Scottsdale, Arizona
  - Clinical Research Center, Encinitas, California
  - AABI Associates Medical Group, Fountain Valley, California
  - William Ebbling, MD Inc, Fresno, California
  - Allergy & Asthma Care Center of So. Cal, Long Beach, California
  - Allergy Research Foundation, Los Angeles, California
  - Southern California Research, Mission Viejo, California
  - Allergy Associates Medical Group Inc, San Diego, California
  - Bensch Research Associates, Stockton, California
  - Storms Clinical Research Institute, Colorado Springs, Colorado
  - Colorado Allergy and Asthma Centers, Denver, Colorado
  - Clinical Research Atlanta, Atlanta, Georgia
  - Atlanta Allergy and Asthma Clinic, Stockbridge, Georgia
  - Clinical Research Atlanta, Stockbridge, Georgia
  - Sneeze, Wheeze and Itch Associates, Normal, Illinois
  - Kansas City Allergy and Asthma, Overland Park, Kansas
  - Northeast Medical Research Associates, North Dartmouth, Massachusetts
  - Clinical Reseacrh Institute, Minneapolis, Minnesota
  - Clinical Research Institute, Plymouth, Minnesota
  - The Clinical Research Center, St Louis, Missouri
  - The Asthma and Allergy Center, Papillion, Nebraska
  - Atlantic Research Center, Ocean City, New Jersey
  - Princeton Center for Clinical Research, Skillman, New Jersey
  - Research Asthma, Sinus and Allergy Centers, Warren Township, New Jersey
  - North Carolina Clinical Research, Raleigh, North Carolina
  - Bernstein Clinical Research Center, Cincinnati, Ohio
  - Allergy and Consultants of NJ/PA, Collegeville, Pennsylvania
  - Allergy and Clinical Immunology Associates, Pittsburgh, Pennsylvania
  - Asthma and Allergy Research Associate, Upland, Pennsylvania
  - National Allergy, Asthma and Urticaria of Charleston, Charleston, South Carolina
  - East Tennesse Center for Clinical Research, Knoxville, Tennessee
  - Allergy and Asthma Associates, Austin, Texas
  - Allergy and Asthma Center of Austin, Austin, Texas
  - AARA Research Center, Dallas, Texas
  - Jane Lee, MD, PA Research Center, Dallas, Texas
  - Central Texas Health Research, New Braunfels, Texas
  - Southwest Allergy and Asthma Center, P.A., San Antonio, Texas
  - Sylvana Research Associates, San Antonio, Texas
  - Intermountain Clinical Research, Draper, Utah

RESULTS

PARTICIPANT FLOW:
Groups:
- MP29-02: azelastine HCl/fluticasone propionate
- Azelastine HCL: active comparator of azelastine HCl
- Fluticasone Propionate: active comparator of fluticasone propionate
- Placebo: placebo control
Period: Overall Study
Arm/Group | MP29-02 | Azelastine HCL | Fluticasone Propionate | Placebo
Started | 193 | 194 | 189 | 200
Completed | 183 | 186 | 180 | 190
Not Completed | 10 | 8 | 9 | 10
Not completed — Adverse Event | 3 | 1 | 1 | 3
Not completed — Lack of Efficacy | 1 | 1 | 0 | 3
Not completed — Lost to Follow-up | 2 | 1 | 0 | 0
Not completed — Protocol Violation | 0 | 1 | 0 | 2
Not completed — Withdrawal by Subject | 1 | 1 | 0 | 0
Not completed — administrative | 3 | 3 | 8 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MP29-02 | Azelastine HCL | Fluticasone Propionate | Placebo | Total
Number analyzed (Participants) | 193 | 194 | 189 | 200 | 776
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 12 | 12 | 14 | 17 | 55
  Between 18 and 65 years | 176 | 178 | 172 | 181 | 707
  >=65 years | 5 | 4 | 3 | 2 | 14
Age Continuous [Mean (Standard Deviation); unit: years] | 38.8 (14.1) | 38.2 (13.5) | 37.0 (13.6) | 37.2 (13.0) | 37.8 (13.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 126 | 128 | 121 | 119 | 494
  Male | 67 | 66 | 68 | 81 | 282
Region of Enrollment [Number; unit: participants]
  United States | 193 | 194 | 189 | 200 | 776

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in 12 Hour Reflective Total Nasal Symptom Score (rTNSS)
Description: change from baseline in 12-hour reflective(how you felt over the previous 12 hours) total nasal symptom score (rTNSS)consisting of nasal congestion,runny nose, itchy nose and sneezing scored twice daily (AM and PM) in diary cards for the entire 14 day study period.
  The measurement scale is 0 to 24.A reduction in symptom severity score is indicated by a negative value.A greater negative score is suggestive of improvement.
Time Frame: day1 to 14 days
Population: Intent-to-Treat(ITT) population includes all subjects who were randomized and had at least one post baseline efficacy observation
Measure: Least Squares Mean (Standard Deviation); unit: units on a scale
Arm/Group | MP29-02 | Azelastine HCL | Fluticasone Propionate | Placebo
Number analyzed (Participants) | 193 | 194 | 189 | 200
units on a scale | -5.5 (5.2) | -4.5 (4.6) | -4.6 (5.1) | -3.0 (3.9)

2. Secondary Outcome: Change From Baseline in 12 Hour Instantaneous Total Nasal Symptom Score (iTNSS)
Description: change from baseline in 12-hour instantaneous ( how do you feel now) total nasal symptom score (iTNSS)consisting of nasal congestion,runny nose, itchy nose and sneezing scored twice daily (AM and PM) in diary cards for the entire 14 day study period.
  The measurement scale is 0 to 24.A reduction in symptom severity score is indicated by a negative value.A greater negative value is suggestive of improvement.
Time Frame: day 1 to14
Population: Intent to Treat (ITT)population includes all subjects who were randomized and had at least one post baseline efficacy observation.
Measure: Least Squares Mean (Standard Deviation); unit: units on a scale
Arm/Group | MP29-02 | Azelastine HCL | Fluticasone Propionate | Placebo
Number analyzed (Participants) | 193 | 193 | 188 | 199
units on a scale | -5.2 (5.3) | -4.2 (4.6) | -4.3 (5.2) | -2.4 (4.2)

3. Secondary Outcome: Change From Baseline in Rhinoconjunctivitis Quality of Life Questionnaire (RQLQ)
Description: adult Rhinoconjunctivitis Quality of Life Questionnaire (RQLQ) scored at day 1(baseline) and at day 14.The scale is measured from a value of 0 to 24. A negative number corresponds to a change from baseline measurement. An increased negative number is suggestive of improvement.
Time Frame: day 1 to day 14
Population: Intent to Treat (ITT) population (18 yrs of age and older) who have had one post baseline efficacy observation
Measure: Least Squares Mean (Standard Deviation); unit: units on a scale
Arm/Group | MP29-02 | Azelastine HCL | Fluticasone Propionate | Placebo
Number analyzed (Participants) | 176 | 172 | 169 | 171
units on a scale | -1.7 (1.3) | -1.4 (1.3) | -1.5 (1.3) | -1.0 (1.3)

ADVERSE EVENTS:
Arm/Group | MP29-02 | Azelastine HCL | Fluticasone Propionate | Placebo
Serious Adverse Events (participants affected / at risk) | 1/193 | 0/194 | 0/189 | 0/200
Other Adverse Events (participants affected / at risk) | 24/193 | 33/194 | 15/189 | 13/200
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MP29-02 (N=193) | Azelastine HCL (N=194) | Fluticasone Propionate (N=189) | Placebo (N=200)
hepatitis C (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — described by investigator as "unlikely related to study drug"
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MP29-02 (N=193) | Azelastine HCL (N=194) | Fluticasone Propionate (N=189) | Placebo (N=200)
headache (Nervous system disorders) | 6 (6) | 4 (4) | 5 (5) | 2 (2)
dysgeusia (Gastrointestinal disorders) | 4 (4) | 14 (14) | 1 (1) | 1 (1)
epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (4) | 3 (5) | 5 (5)
mucosal erosion (General disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (4) | 5 (5) | 2 (2)
cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
upper respiratory tract infection (Infections and infestations) | 1 (1) | 2 (2) | 1 (1) | 1 (1)
nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
nasopharyingitis (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigators participating in multicenter studies must agree not to present data gathered individually or by a subgroup of centers before the full, initial publication, unless this has been agreed to by all other investigators and Meda Pharmaceuticals.

Meda Pharmaceuticals requests that it receive copies of any intended communication reasonably in advance (at least 15 working days for an abstract or oral presentation and 45 working days for a manuscript)